CLINICAL TRIAL: NCT06188832
Title: Efficacy of Dietary Fiber Supplementation (Soloways) in Patients With Specific Genetic Polymorphisms
Acronym: SOLFIBERGP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center of New Medical Technologies (Other); Triangel Scientific (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SW003
Record Dates: First submitted 2023-12-07; First posted 2024-01-03 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: obesity; supplements; body mass index; overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — (1-6)-alpha-glucomannan; Inulin; Psyllium

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber Supplementation (Experimental): The active powder contained 1g glucomannan, 1g inulin, and 3g psyllium per bag.
  Interventions: Dietary Supplement: glucomannan, inulin, and psyllium
- Placebo group (Placebo Comparator): The placebo powder composed of maltodextrin and rice flour, carefully selected to mimic the texture and volume of the active powder without providing any active dietary fiber
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: glucomannan, inulin, and psyllium — the subjects recieved fiber supplement containing glucomannan, inulin, and psyllium
  Arms: Fiber Supplementation
Other: placebo — the subjects recieved placebo
  Arms: Placebo group

SUMMARY:
This randomized, double-blind, placebo-controlled trial assessed the impact of a dietary fiber supplement (glucomannan, inulin, and psyllium) on weight and metabolic parameters in individuals with obesity-related genetic polymorphisms (FTO, MC4R, LEP, LEPR). Participants were adults aged 18-65 with a BMI ≥ 25 and confirmed genetic predispositions. The study, involving 216 participants (108 per group), ran over 12 weeks with assessments at 0, 4, 8, and 12 weeks. Primary outcome was Body-weight change in %. The study aimed to clarify the role of fiber supplements in genetically predisposed obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed presence of one or more specified gene polymorphisms (FTO, MC4R, LEP, LEPR).
* Overweight or obese status (BMI ≥ 25).

Exclusion Criteria:

- BMI < 25

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Body-weight change in % | 180 days

SECONDARY OUTCOMES:
body-weight reduction ≥5% | 180 days
body-weight reduc-tion ≥10% | 180 days
Body weight in kg | 180 days
Body mass index change in % | 180 days
Fat mass change in % | 180 days
Systolic blood pressure in mmHg | 180 days
Fat-free mass change in kg | 180 days
Visceral fat rating change from baseline | 180 days
Diastolic blood pressure in mmHg | 180 days
Total cholesterol ratio | 180 days
LDL-C ratio | 180 days
HDL-C ratio | 180 days
Triglycerides ratio | 180 days
hsCRP ratio | 180 days
Fasting plasma glucose mmol/l | 180 days
Side effects % | 180 days
  any side effects or adverse events reported by subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Center of New Medical Technologies, Novosibirsk, Novosibisk Region, Russia

REFERENCES:
- [Result] Pokushalov E, Ponomarenko A, Garcia C, Pak I, Shrainer E, Seryakova M, Johnson M, Miller R. The Impact of Glucomannan, Inulin, and Psyllium Supplementation (SolowaysTM) on Weight Loss in Adults with FTO, LEP, LEPR, and MC4R Polymorphisms: A Randomized, Double-Blind, Placebo-Controlled Trial. Nutrients. 2024 Feb 17;16(4):557. doi: 10.3390/nu16040557. PMID 38398881
- See also: 10.3390/nu16040557 — https://pubmed.ncbi.nlm.nih.gov/38398881/